CLINICAL TRIAL: NCT01850407
Title: Preparing Caregivers for the Child Sexual Abuse Examination: Are Informational Leaflets Helpful?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 07.02.054
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Child Sexual Abuse, Suspected
Keywords: Lack of Preparation for Abused Children during Medical Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Education Counseling (No Intervention): Education of caregivers to counter lack of Preparedness for Children Undergoing Sexual Abuse Medical Examination
  Interventions: Behavioral: Education Counseling

INTERVENTIONS:
Behavioral: Education Counseling

SUMMARY:
Children are typically inadequately prepared for the sexual abuse medical examination. Caregivers report lack of examination knowledge as a barrier to preparing their children. The purpose of this study was to determine if informational leaflets provided prior to the examination are helpful to caregivers in preparing their children.

ELIGIBILITY:
Inclusion Criteria:

* consecutive caregivers accompanying children for scheduled sexual abuse medical examination

Exclusion Criteria:

* Lack of consent
* Failure to complete study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-08; Primary Completion 2007-12 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To determine the helpfulness of informational leaflets in preparing caregivers for the child sex abuse examination | one month
  [The study] undertook a prospective study of consecutive caregivers accompanying children for a scheduled sexual abuse medical examination. Prior to the appointment, caregivers were mailed information leaflets (in English and Spanish) about how to prepare their children for the exam. Caregivers completed pre and post exam surveys and the State-Trait Anxiety Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Agrawal, MD, Principal Investigator — Hackensack Meridian Health